CLINICAL TRIAL: NCT02203825
Title: A Phase 1 Study of Chimeric Antigen Receptor Modified T-cells Targeting NKG2D-Ligands in Patients With Acute Myeloid Leukemia (AML)/Advanced Myelodysplastic Syndrome (MDS-RAEB) and Multiple Myeloma.
Brief Title: Safety Study of Chimeric Antigen Receptor Modified T-cells Targeting NKG2D-Ligands
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celyad Oncology SA (Industry)
Collaborators: Dana-Farber Cancer Institute (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM-14-001; 5R44HL099217-03 (NIH)
Record Dates: First submitted 2014-07-25; First posted 2014-07-30 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Multiple Myeloma
Keywords: Acute Myeloid Leukemia; NKG2D; Multiple Myeloma; Cell Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CM-CS1 T-cell infusion (Experimental): The treatment will consist of a single infusion of CM-CS1 cells.
  The following dose levels will be evaluated:
  Cohort 1: 1x 10^6 CM-CS1 T-cells Cohort 2: 3x 10^6 CM-CS1 T-cells Cohort 3: 1x 10^7 CM-CS1 T-cells Cohort 4: 3x 10^7 CM-CS1 T-cells
  Interventions: Biological: CM-CS1 T-cell infusion

INTERVENTIONS:
Biological: CM-CS1 T-cell infusion — Each patient will receive a single dose of CM-CS1 T-cells by intravenous infusion.

SUMMARY:
This Phase I clinical trial is evaluating chimeric-antigen receptor (CAR) T-cells (CM-CS1 T cells) which recognize NKG2D-ligands on the surface of cancer cells. This study evaluates the safety and feasibility of administering a single intravenous dose of CM-CS1 CAR T-cells to patients with AML, MDS-RAEB and Multiple Myeloma.

DETAILED DESCRIPTION:
This is a study for patients with AML or MDS-RAEB that is not in remission and for which there are no reasonable standard treatment options and for patients with relapsed/refractory multiple myeloma with progressive disease.

In this study, the participant's white blood cells (T-cells) will be collected and modified such that the T-cells are able to recognize specific molecules (called NKG2D-ligands), that are expressed on the surface of cancer cells in these diseases. This modification is a genetic change to the T-cells. The modified T cells, called CM-CS1 T-cells, are then given back to the participant by a single intravenous infusion. In this study, participants will not receive any chemotherapy prior to infusion of the CM-CS1 T-cells.

The study will evaluate whether it is safe and feasible to administer CM-CS1 T-cells to participants with AML/MDS-RAEB and multiple myeloma. It will also evaluate whether the CM-CS1 T-cells have a beneficial effect against the cancer cells. Another goal of the study is to learn more about the persistence and function of the CM-CS1 T-cells in the body.

Participants will be followed very closely during the first month after infusion. They are required to remain within 50 miles of Brigham and Women's Hospital (Boston, MA) for 10 days after the infusion and will be followed three times per week for the first 21 days and at day 28. Subsequently, participants will be followed monthly until 6 months after infusion, every 3 months until 15 months after infusion and at 24 months after infusion. Because this study involves gene transfer, participants will be followed yearly for up to 15 years.

ELIGIBILITY:
General eligibility criteria:

* ECOG performance status 0 or 1.Patients with multiple myeloma who have an ECOG performance status of 2 based on peripheral neuropathy from prior therapies are eligible.
* Ability to understand and the willingness to sign a written informed consent document.
* Pathological confirmation of AML, MDS-RAEB or Multiple myeloma.
* Agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of CM-CS1 CART-cell administration.
* Ability to adhere with the study visit schedule and other protocol procedures.
* Willingness to remain within a 50 mile radius of Brigham Women's Hospital during the initial 10 days following CM-CS1 infusion

Disease specific eligibility criteria for patients with AML, MDS-RAEB:

* Pathological confirmation of AML, MDS-RAEB according to WHO classification (CMML is excluded) that is not in remission (defined as >5% blasts in bone marrow or peripheral blood) and for which there are no reasonable standard treatment options.
* No known or suspected CNS disease. A neurologic exam is required and signs or symptoms suggestive of potential CNS disease require CNS imaging.
* Disease status deemed not to require additional therapy for at least 4 weeks from enrollment.
* Life expectancy of greater than 4 weeks.
* Participants must have satisfactory organ function as defined below:

  1. Total bilirubin ≤2.0 × institutional upper limit of normal (Except for subjects with known Gilbert's syndrome)
  2. AST(SGOT)/ALT(SGPT) ≤3 × institutional upper limit of normal
  3. Creatinine ≤ 2.0 mg/dL

Disease specific eligibility criteria for patients with multiple myeloma:

* Diagnosis of active multiple myeloma according to the International Myeloma Working Group diagnostic criteria.
* Relapsed or relapsed/refractory multiple myeloma with progressive disease
* Presence of measurable disease as defined as one or more of the following:

  1. Serum M-protein >0.5g/dl
  2. Urine M-protein > 200mg/24hr
  3. Serum FLC assay: involved FLC level > 10mg/dl with abnormal serum FLC ratio
  4. Measurable plasmocytoma in non-secretory patients.
* Previous treatment with both an immunomodulator and a proteosome inhibitor therapy
* Life expectancy of greater than 12 weeks
* No known or suspected CNS involvement. A neurologic exam is required and signs or symptoms of potential CNS involvement require CNS imaging. Peripheral neuropathy is acceptable.
* Participants must have satisfactory organ and marrow function as defined below:

  1. Absolute neutrophil count > 500/mcL. Screening ANC should be independent of G-CSF and GM-CSF support for at least 1 week and of pegylated G-CSF for at least 2 weeks
  2. Platelets >20,000/mcL. Subjects may receive platelet transfusions, if clinically indicated, in accordance with institutional guidelines.
  3. Total bilirubin ≤2.0 × institutional upper limit of normal. (Except patients with known Gilbert's syndrome)
  4. AST(SGOT)/ALT(SGPT) ≤3 × institutional upper limit of normal
  5. Creatinine ≤ 2.0 mg/dL

Exclusion Criteria:

* Participants who have received chemotherapy or radiotherapy within 3 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier.
* Concurrent systemic steroid or other immunosuppressive therapy.
* Participants who are concurrently receiving any other investigational agents, or have received another investigational agent within 3 weeks before enrollment.
* Participants who have received prior allogeneic stem cell transplantation, gene therapy, or adoptive T-cell therapy.
* Active infections necessitating use of treatment antibiotics/antivirals during the screening period (prophylaxis is acceptable) or evidence of an active communicable infectious disease.
* Participants who underwent major surgery within 4 weeks before day 0 of planned CM-CS1 T-cell infusion (this does not include placement of vascular access device or tumor biopsies).
* Participants with any known history of primary immunodeficiency.
* History of allergic reactions or hypersensitivity attributed to Human serum albumin or Plasma-lyte A.
* Uncontrolled intercurrent illness or serious uncontrolled medical disorder
* Pregnancy or breastfeeding
* Known HIV-positive participants are ineligible because the effect of transducing HIV-infected lymphocytes with the chimeric NKG2D- transgene on the disease course is unknown.
* Clinically relevant active infection including active hepatitis B or C or any other concurrent disease which in the judgment of the Investigator would make the subject inappropriate for enrollment on this study.
* Active autoimmune disease
* History of a malignancy other than one of the malignancies in this study with exception of the following circumstances:

  1. Patients with a history of malignancy who have been adequately treated and have been disease-free for at least 2 years are not excluded.
  2. Patients with adequately treated active non-invasive cancers (such as non-melanomatous skin cancer or in-situ bladder, cervical and breast cancers) are not excluded.
* Unwillingness to use an effective contraceptive method during the study and at least 4 months after administration of CM-CS1 T-cells unless subject is naturally infertile.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility of intravenous administration of CM-CS1 T-cells. | 24 months
  Safety will be defined by the occurence of study-related serious and non-serious adverse events.
  Feasibility will be defined by the frequency of subjects enrolled who do not receive CM-CS1 T-cells.

SECONDARY OUTCOMES:
Clinical and biologic responses | 24 months
  Clinical anti-tumor effect by standard criteria Progression-Free survival Persistence and function of CM-CS1 T-cells

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Nikiforow, MD; PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Murad JM, Baumeister SH, Werner L, Daley H, Trebeden-Negre H, Reder J, Sentman CL, Gilham D, Lehmann F, Snykers S, Sentman ML, Wade T, Schmucker A, Fanger MW, Dranoff G, Ritz J, Nikiforow S. Manufacturing development and clinical production of NKG2D chimeric antigen receptor-expressing T cells for autologous adoptive cell therapy. Cytotherapy. 2018 Jul;20(7):952-963. doi: 10.1016/j.jcyt.2018.05.001. Epub 2018 Jun 29. PMID 30180944
- See also: Sponsor — http://www.celyad.com